CLINICAL TRIAL: NCT01886118
Title: A Randomized Trial Evaluating Autologous Endometrial Co-Culture Versus Conventional Medium in the Treatment of Infertility
Brief Title: A Trial Evaluating Autologous Endometrial Co-Culture Versus Conventional Medium in the Treatment of Infertility
Acronym: OvoGEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Ovo (Industry)
Collaborators: Genevrier Laboratories (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OVO-12-24
Record Dates: First submitted 2013-01-03; First posted 2013-06-25 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
Keywords: In vitro fertilization; Autologous Endometrial Co-Culture
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous Endometrial Co-Culture (Experimental): The embryos will be transferred to Endocell co-culture media for Autologous Endometrial Co-Culture between day 2 and day 5.
  Interventions: Procedure: Endometrial biopsy; Other: Autologous Endometrial Co-Culture
- Conventional media culture (Active Comparator): Patients in this arm will have their embryos cultured in conventional media
  Interventions: Procedure: Endometrial biopsy; Other: Conventional media culture

INTERVENTIONS:
Procedure: Endometrial biopsy — A luteal phase endometrial biopsy will be performed in the cycle prior to the patient's In Vitro Fertilization stimulation cycle using a standard Pipelle Endometrial Suction curette in all participants between days ovulation+5 and ovulation+7 of the cycle preceding the stimulation cycle
Other: Autologous Endometrial Co-Culture — embryos will be transferred to Endocell co-culture media for Autologous Endometrial Co-Culture between day 2 and day 5
  Arms: Autologous Endometrial Co-Culture
Other: Conventional media culture — embryos are cultured in conventional media
  Arms: Conventional media culture

SUMMARY:
One of the main factors in the success of in-vitro fertilization is the quality of the environment of the embryo. In contrast to maternal age, the environment in which the embryo develops is a modifiable factor. Many techniques, such as assisted hatching and perfecting culture media have been attempted in order to reproduce as much as possible the natural, physiological environment of the mother for the embryo in in-vitro fertilization. However, the different new culture media used are devoid of growth factors normally secreted by uterine cells that enhance the interaction between the embryo and its environment.

Because the endometrial lining of the uterus secretes many different cytokines necessary for growth of the embryo, a new procedure has been developed to mimic the natural environment of the growing embryo using autologous (patient's own) endometrial cells in co-culture with the embryo. Endocell, a product developed by Genévrier Laboratories, received commercial authorization in France in 2011. It is the only system of autologous embryo-endometrium co-culture available on the actual market. The process consists of developing the embryo on a monolayer of the patient's own endometrial cells in order to favor its growth until the blastocyst stage (day 5) and to improve its implantation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing In Vitro Fertilization (IVF) or IVF/Intra Cytoplasmic Sperm Injection (ICSI) at OVO clinic
* Having a prescription of a long, short or an antagonist IVF protocols using both urinary and synthetic gonadotropins
* Having a single embryo transfer
* Regular menstrual cycles
* Basal follicle stimulating hormone levels less than 10 IU/l within 6 months prior to entering the study
* anti-mullerian hormone more than 1 ng/ml measured within a year
* Normal sonohysterogram or hysteroscopy done within the last 2 years
* Previously undergone a maximum of 3 IVF cycles
* Documented negative serology tests within 1 year prior recruitment for: Hepatitis B, Syphilis, HIV based on Health Canada recommendations for treatment in an IVF laboratory.

Exclusion Criteria:

* Amenorrhea
* Anovulatory cycles
* Polycystic Ovarian syndrome
* Chronic endometritis
* Severe endometriosis
* Hydrosalpinx
* Uterine synechia or Asherman's syndrome
* Submucosal uterine fibroids or intra-cavitary polyps greater than 1cm
* Uterine anomalies
* Use of anticoagulants
* Secretory Azoospermia

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pregnancy rates | 7 weeks
  Confirmed clinical pregnancy with positive fetal heart on the day of viability ultrasound

SECONDARY OUTCOMES:
Embryo quality | 5 days
  The number of cells and the grade of the embryos will be assess throughout their development.
Blastulation rate | 5 days
  Percentage of embryos that develops into blastocyst compared to the total number of embryos in culture
Cumulative pregnancy rate with frozen embryos | 5 years
  Pregnancy rate per patient including all transfer with frozen embryos

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada